CLINICAL TRIAL: NCT06582082
Title: Digital Health Integration With Pulmonary Rehabilitation on Ventilatory, Cognitive and Physical Functions in Patients With Chronic Obstructive Lung Disease
Brief Title: Digital Health Integration With Pulmonary Rehabilitation on Patients With Chronic Obstructive Lung Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa mahmoud elsayed mahmoud, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: P.T.REC/012/005239
Record Dates: First submitted 2024-08-28; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulmonary rehabilitation (Experimental): The study group will receive pulmonary rehabilitation
  Interventions: Other: pulmonary rehabilitation
- lip breathing (Active Comparator): the control group will stick to pursed lip breathing only
  Interventions: Other: pursed lip breathing

INTERVENTIONS:
Other: pulmonary rehabilitation — The study group will receive pulmonary rehabilitation
  Arms: pulmonary rehabilitation
Other: pursed lip breathing — the control group will stick to pursed lip breathing only
  Arms: lip breathing

SUMMARY:
It is an interventional study in which 60 COPD patients estimated to enrol according to random allocation and divided into two groups. The study group will receive pulmonary rehabilitation while the control group will stick to pursed lip breathing only.

Pulmonary function (FEV1, FVC, FEV1/FVC), cognitive function by mini mental state examination, physical function by physical tests also, physical activity and sleep by google fit app and vital signs by using different mobile apps. measurements will be evaluated before initiation of the interventions and 12 weeks thereafter.

DETAILED DESCRIPTION:
PURPOSE:

to evaluate the efficacy of Digital Health Integration with pulmonary rehabilitation on ventilatory, cognitive and physical functions in patients with chronic obstructive lung disease.

BACKGROUND:

chronic obstructive pulmonary diseases are conditions characterized by a variable progression. Some individuals experience longer asymptomatic periods while others acute worsening periods and/or exacerbations triggered by symptom multiplication factors. Medications are adjusted to the patients' respiratory function, self-assessment of health and emerging certain physical changes. A more effective treatment may be applied by real-time data registered during the patient's everyday life Effective, safe, accessible, and engaging digital healthcare solutions which are able to be integrated into global healthcare systems may play a role in helping to meet this demand in COPD care needs. Digital interventions are unrestricted by individual practices or healthcare systems and come in a range of forms, including: synchronous applications (apps) which provide real-time video conferencing or telephone calls; asynchronous solutions such as emails, smartphone messages, or notifications; remote monitoring or recording devices, such as traditional telehealth interventions; information providing devices; and modern multi-tooled digital health apps which can facilitate behavioural changes and self-management..

HYPOTHESES:

Digital Health Integration with pulmonary rehabilitation has no effect on ventilatory, cognitive and physical functions in patients with chronic obstructive lung disease.

RESEARCH QUESTION:

Does Digital Health Integration with pulmonary rehabilitation influence ventilatory, cognitive and physical functions in patients with chronic obstructive lung disease?

ELIGIBILITY:
Inclusion Criteria:

* All gender COPD patients
* Age will be 55-65 years.
* Moderate to severe COPD patients
* emphysema on CT scan (HU ≥ - 900)
* There FEV1 will be less than 80% predicted
* Class II obesity (BMI of 35 to < 40)
* Medically stable
* greater than 10 pack-year smoking history

Exclusion Criteria:

* Very severe COPD - Lung cancer
* Lung resection - Lung fibrosis
* Heart failure - Cognitive disorders that affect the device application
* Musculoskeletal or neurological disorders that interfere with exercise program
* requiring invasive or non-invasive positive pressure ventilation
* inability to speak in complete sentences due to breathlessness
* suspected elevated intracranial pressure - hemodynamic instability
* recent facial, oral, or skull surgery
* active hemoptysis (more than two tablespoons of frank blood per day)
* pneumothorax - failure to comply with the research protocol.
* uncontrolled hypertension, or other concomitant respiratory diseases
* participate at any research or pulmonary rehabilitation program during the period of this study.
* imaging changes of lung disease such as occupancy, exudation and interstitial changes on CT scan.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
pulmonary function | 12 weeks
  Pulmonary function test will be carried out by SPIROVIT SP-1 spirometer to determine FVC, FEV1, FEV1/FVC. Subjects will remain in the straight sitting or standing position throughout the test, and a nose clip will be tightly attached to the nostrils, allowing no air to escape during the test. A mouthpiece will be placed at least two centimeters into the subject's mouth, with lips closed around it.

SECONDARY OUTCOMES:
cognitive function | 12 weeks
  A Mini-Mental State Examination (MMSE) is a set of 11 questions. It's used by to check for cognitive impairment. The test takes about 5 to 10 minutes. The top score for the MMSE is 30 - a score of 25 or higher is said to be normal.
physical activity | 12 weeks
  The Google Fit® is an open platform developed by Google Inc., which allows the users to control their fitness data. It is also available as a free application for smartphones, which works with versions above 4.0 in Android systems. The Google Fit® consists of a set of high level sensors, such as an accelerometer, a gyroscope, and a GPS system which can detect changes in position (for example, moving from sitting to standing), various types of movement (walking, cycling, and others), several kinds of data (number of steps, walked distance, heart rate, and others), and different bouts of activity (time of each bout) ( Google Developers, 2016
  ).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
sharing study protocol with other researchers
Supporting Information: Study Protocol
Time Frame: two years
Access Criteria: up on appropriate request of corresponding author
URL: http://www.ekb.com